CLINICAL TRIAL: NCT06419218
Title: Evaluating a Marketing Campaign to Increase Participation in School Meals
Brief Title: Increasing School Meal Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Anna Grummon, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 75335
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Nutrition, Healthy
Keywords: health; nutrition; children; parent perceptions; school lunch; school breakfast; food access

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator and data analyst will not be aware of participants' assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School meal messages (Experimental): Participants will view messages focused on the benefits of children eating school meals, using text and images developed based on parent interviews. Participants will view a total of 10 messages.
  Interventions: Behavioral: School meal messages
- Control (neutral) messages (Active Comparator): Participants will view messages focused on the benefits of children reading. Messages will be matched in length to the experimental messages. Participants will view a total of 10 messages.
  Interventions: Behavioral: Control (neutral) messages

INTERVENTIONS:
Behavioral: School meal messages — Messages focused on the benefits of children consuming school lunch and breakfast, using text and images developed based on parent interviews. Participants will view a total of 10 messages.
  Arms: School meal messages
Behavioral: Control (neutral) messages — Control messages approximately matched to the intervention messages on length and design, but discussing a neutral topic unrelated to school meals (reading). Participants will view a total of 10 messages.
  Arms: Control (neutral) messages

SUMMARY:
This study aims to determine whether an online marketing campaign increases children's school meal participation. Parents whose children do not currently eat school meals frequently will be exposed to messages designed to encourage their children's increased participation in school meals.

DETAILED DESCRIPTION:
In this 6-week-long online randomized controlled trial, participants will be randomized to one of two arms: 1) Control (neutral) messages or 2) Messages designed to increase school meal participation. In each arm, participants will join private Facebook groups corresponding to their study arm. The study team will post campaign messages to these groups. Participants will answer online survey questions before and after the study on their attitudes about school meals and their child's participation in school meals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Parent of a child attending a public school in grades 1-5
* Resides in one of the following states: California, Colorado, Maine, Minnesota, Michigan, Massachusetts, New Mexico, Vermont
* Has internet access
* Has a Facebook account
* Child consumes 3 or fewer school lunches per week or 3 or fewer school breakfasts per week

Exclusion Criteria:

* Younger than 18 years old
* Does not have a child attending a public school in grades 1-5
* Resides out of one of the following states: California, Colorado, Maine, Minnesota, Michigan, Massachusetts, New Mexico, Vermont
* Does not have internet access
* Does not have a Facebook account
* Child consumes more than 3 school lunches per week and more than 3 school breakfasts per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 832 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Children's consumption of school lunches | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental report of the usual number of days per week their child ate school lunch during the past month. Assessed with 1 item: "Thinking about the last month, how many days a week did your child usually eat school lunch?" This item will be scored on a 6-point scale from "0 days per week" (0) to "5 days per week" (5).
Children's consumption of school breakfasts | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental report of the usual number of days per week their child ate school breakfast during the past month. Assessed with 1 item: Thinking about the last month, how many days a week did your child usually eat school breakfast?" This item will be scored on a 6-point scale from "0 days per week" (0) to "5 days per week" (5).

SECONDARY OUTCOMES:
Noticing the school meal campaign | Collected in a ~10 minute survey at 6 weeks.
  Parental report of whether they noticed the school meal campaign. Assessed with 1 item: "In the last 6 weeks, have you seen any messages or advertising on Facebook encouraging children to eat school lunch or school breakfast?" Response options are "yes" (1) and "no" (0).
Number of school meals campaign topics recognized | Collected in a ~10 minute survey at 6 weeks.
  Parental report of the number of topics they recognize having seen in messages about school meals. Assessed with 1 item: "Which of these topics did the messages discuss, if any? Check all that apply." Response options list 8 topics plus options for "none of these" and "not sure." Number of topics recognized will be calculated as the sum of all topics that parents indicate they have seen. Those who answer, "none of these" and "not sure" will be coded as recognizing 0 topics. Those who report not noticing the school meal marketing campaign will be coded as recognizing 0 topics.
Frequency of reading campaign messages | Collected in a ~10 minute survey at 6 weeks.
  Parental report of the frequency with which they read their assigned campaign messages. Assessed with 1 item: "In the past month, how often did you read these messages?" This item will be scored on a 5 point scale ranging from "Never or less than 1 time per week" (1) to "Every day or more often" (5).
Social interactions about campaign | Collected in a ~10 minute survey at 6 weeks.
  Parental report of the frequency with which they talked to others about their assigned campaign messages. Assessed with 1 item: "In the last month, how often did you talk to others about these messages?" This item will be scored on a 5 point scale ranging from "Never or less than 1 time per week" (1) to "Every day or more often" (5).
Social interactions about school meals | Collected in a ~10 minute survey at 6 weeks.
  Parental report of the frequency with which they talked to others about school meals. Assessed with 3 items (e.g., "In the last month, how often did you talk to others about school meals?"). Response options are on a 5-point scale ranging from "Never or less than 1 time per week" (1) to "Every day or more often" (5). Responses to the 3 items will be averaged to create a mean score.
Perceived benefits of school lunch | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental report of the benefits of their child consuming school lunch. Assessed with 8 items (e.g., "My child eating school lunch helps my child do well in school"). Response options are on a 5-point scale ranging from "Strongly disagree" (1) to "Strongly agree" (5). Responses to the 8 items will be averaged to create a mean score.
Perceived benefits of school breakfast | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental report of the benefits of their child consuming school breakfast. Assessed with 8 items (e.g., "My child eating school breakfast helps my child do well in school"). Response options are on a 5-point scale ranging from "Strongly disagree" (1) to "Strongly agree" (5). Responses to the 8 items will be averaged to create a mean score.
Knowledge that school lunch is free | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental knowledge that lunches served at their child's school are free to all students. Assessed with 1 item: "Are school lunches free for all students at your child's school?" Response options "yes" (coded as 1) and "no" or "not sure" (both coded as 0).
Knowledge that school breakfast is free | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental knowledge that breakfasts served at their child's school are free to all students. Assessed with 1 item: "Are school breakfasts free for all students at your child's school?" Response options "yes" (coded as 1) and "no" or "not sure" (both coded as 0).
Perceived healthfulness of school lunch | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental perception of the healthfulness of the lunches served at their child's school. Assessed with 1 item: "How healthy or unhealthy are the school lunches at your child's school?" Response options are on a 5-point scale ranging from "Very unhealthy" (1) to "Very healthy" (5).
Perceived healthfulness of school breakfast | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental perception of the healthfulness of the breakfasts served at their child's school. Assessed with 1 item: "How healthy or unhealthy are the school breakfasts at your child's school?" Response options are on a 5-point scale ranging from "Very unhealthy" (1) to "Very healthy" (5).
Intentions to encourage their children's consumption of school lunch | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental report of the likelihood of encouraging their child to eat school lunch in the next month. Assessed with 1 item: "In the next month, how likely are you to encourage your child to eat school lunch?" Response options are on a 5-point scale ranging from "Not at all likely" (1) to "Extremely likely" (5).
Intentions to encourage their children's consumption of school breakfast | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental report of the likelihood of encouraging their child to eat school breakfast in the next month. Assessed with 1 item: "In the next month, how likely are you to encourage your child to eat school breakfast?" Response options are on a 5-point scale ranging from "Not at all likely" (1) to "Extremely likely" (5).
Barriers to children's school lunch consumption | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental report of the barriers preventing their child from eating school lunch. Assessed with 1 item: "What are some reasons that your child doesn't eat school lunch more often? Check all of the reasons that apply." Response options list 15 reasons plus "NA - my child eats school lunch every day or almost every day" and a free response option for "other." Total number of barriers selected will be summed. Those who report "NA - my child eats school lunch every day or almost every day" will be coded as having 0 barriers.
Barriers to children's school breakfast consumption | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental report of the barriers preventing their child from eating school breakfast. Assessed with 1 item: "What are some reasons that your child doesn't eat school breakfast more often? Check all of the reasons that apply." Response options list 16 reasons plus "NA - my child eats school breakfast every day or almost every day" and a free response option for "other." Total number of barriers selected will be summed. Those who report "NA - my child eats school breakfast every day or almost every day" will be coded as having 0 barriers.
Household food insecurity | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental report of household food insecurity. Assessed with 6 items (e.g., "In the last month, were you ever hungry but didn't eat because there wasn't enough money for food?") Response options include "no" or "yes"; "never true", "sometimes true", or "often true"; "only 1 or 2 days," "some days but not every day," or "almost every day." Responses of "often" or "sometimes" and "yes" are coded as affirmative (yes). Likewise, responses of "almost every day" and "some days but not every day" are coded as affirmative (yes). The sum of affirmative responses to the six questions in the module is the household's raw score on the scale.
  Household food security status is assigned as follows:
  Raw score 0-1-High or marginal food security Raw score 2-4-Low food security Raw score 5-6-Very low food security Analyses will dichotomize households into those with high or marginal food security and those with low or very low food security.
Child food insecurity | Collected in a ~10 minute survey at baseline and again at 6 weeks.
  Parental report of child food insecurity. Assessed with 8 items (e.g., "In the last month, did you ever cut the size of your child's meals because there wasn't enough money for food?") Response options include "no" or "yes"; "never true", "sometimes true", or "often true"; "only 1 or 2 days," "some days but not every day," or "almost every day." Responses of "often" or "sometimes" and "yes" are coded as affirmative (yes). Responses of "almost every day" and "some days but not every day" are coded as affirmative (yes). The sum of affirmative responses to the 8 questions in the module is the child's raw score on the scale.
  Child food security status is assigned as follows:
  Raw score 0-1-High or marginal food security among children; Raw score 2-4-Low food security among children; Raw score 5-8-Very low food security among children Analyses will dichotomize households into those with children with high or marginal food security or children with low or very low food security.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Grummon, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Stanford School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to post de-identified raw data from the surveys to a public repository.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: We plan to post de-identified raw data from the surveys to a public repository upon publication of papers arising from the study.
Access Criteria: These materials will be posted publicly; researchers will be free to download them.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT06419218/Prot_SAP_000.pdf